CLINICAL TRIAL: NCT02509065
Title: The Set-Point Study: Evaluating Effects of Changing Glucose Target on Bionic Pancreas Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001260
Record Dates: First submitted 2015-07-22; First posted 2015-07-27 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: bionic pancreas; artificial pancreas; insulin; glucagon; continuous glucose monitor (CGM); insulin pump; outpatient
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Masking Description: Some of the study arms are double blinded: the 110 mg/dl and 130 mg/dl set point configurations of the bionic pancreas are double blinded, so neither the patient nor the study team know if they are using the bihormonal bionic pancreas or insulin only bionic pancreas
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Usual Care (Active Comparator): Comparator week to all closed-loop control, utilizing usual diabetes care and the subject's own insulin pump.
  Interventions: Other: Usual Care
- 145 mg/dl Set Point - insulin only (Experimental): Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 145 mg/dl and using only an insulin pump.
  Interventions: Device: Bionic Pancreas
- 130 mg/dl Set Point - insulin only (Experimental): Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 130 mg/dl and using only an insulin pump. This arm is for subjects with type 1 diabetes only. This arm is double blinded; neither the subject nor the study team know if it is insulin only or bihormonal.
  Interventions: Device: Bionic Pancreas
- 130 mg/dl Set Point - bihormonal (Experimental): Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 130 mg/dl using both an insulin and a glucagon pump. This arm is double blinded; neither the subject nor the study team know if it is insulin only or bihormonal.
  Interventions: Device: Bionic Pancreas
- 115 mg/dl Set Point - bihormonal (Experimental): Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 115 mg/dl using both an insulin and a glucagon pump.
  Interventions: Device: Bionic Pancreas
- 100 mg/dl Set Point - bihormonal (Experimental): Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 100 mg/dl using both an insulin and a glucagon pump.
  Interventions: Device: Bionic Pancreas
- 110 mg/dl Set Point - insulin only (Experimental): Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 110 mg/dl and using only an insulin pump. This arm is double blinded; neither the subject nor the study team know if it is insulin only or bihormonal.
  Interventions: Device: Bionic Pancreas
- 110 mg/dl Set Point - bihormonal (Experimental): Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 110 mg/dl using both an insulin and a glucagon pump. This arm is double blinded; neither the subject nor the study team know if it is insulin only or bihormonal.
  Interventions: Device: Bionic Pancreas
- 120 mg/dl Set Point - insulin only (Experimental): Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 120 mg/dl and using only an insulin pump.
  Interventions: Device: Bionic Pancreas

INTERVENTIONS:
Device: Bionic Pancreas — Participant wears the bionic pancreas, including an insulin and/or glucagon pump depending on which arm they are in. The 100 mg/dl arm for type 1 diabetes patients will deliver insulin and glucagon. The 100 mg/dl arm for type 2 diabetes patients will deliver just insulin. The 115 mg/dl arm will deliver insulin and glucagon. The 120 mg/dl arm will deliver just insulin. The 145 mg/dl arm will deliver just insulin. The 130 mg/dl and 110 mg/dl arms will deliver insulin and placebo, or insulin and glucagon, and will be double blinded.
  Arms: 100 mg/dl Set Point - bihormonal; 110 mg/dl Set Point - bihormonal; 110 mg/dl Set Point - insulin only; 115 mg/dl Set Point - bihormonal; 120 mg/dl Set Point - insulin only; 130 mg/dl Set Point - bihormonal; 130 mg/dl Set Point - insulin only; 145 mg/dl Set Point - insulin only
Other: Usual Care — Participant cares for their diabetes according to their usual practice, with blinded CGM monitoring. No medication will be administered by the study in this intervention.
  Arms: Usual Care

SUMMARY:
The current study is designed to determine the effect on mean glucose, hypoglycemia, glucagon usage, and insulin usage of adjusting upward the glucose target of the bi-hormonal bionic pancreas, and determine whether there is a target at which adequate glycemic control is achieved by an insulin-only bionic pancreas with minimal hypoglycemia.

DETAILED DESCRIPTION:
We have two specific aims:

Aim 1 is to conduct an outpatient study testing multiple configurations of the bionic pancreas in 24 adult subjects with type 1 diabetes in a random cross-over study versus usual care with an insulin pump. These bionic pancreas configurations include the insulin only BP at 145 mg/dl set point, 130 mg/dl set point, 120 mg/dl set point and 110 mg/dl set point and the bihormonal BP at 130 mg/dl set point, 115 mg/dl set point and 110 mg/dl set point. These arms are all compared to usual care.

Aim 2 is to evaluate the incremental utility of glucagon in the context of automated insulin delivery by the bionic pancreas in preventing hypoglycemia during exercise in the fasted state. The 130 mg/dl set points and 110 mg/dl set points also participate in this fasted exercise visit. These two set points are double blinded, so neither the subjects nor the study staff are aware which arm is bihormonal and which arm is insulin only.

ELIGIBILITY:
Inclusion Criteria:

Type 1 Diabetes Subjects: Age ≥ 18 years and have had clinical type 1 diabetes for at least one year, and managed using an insulin pump for ≥ 6 months Type 2 Diabetes subjects: Age ≥ 18 years and have type 2 diabetes managed with rapid acting insulin in an insulin pump, or multiple daily injections including both long acting and short acting insulin

* Prescription medication regimen stable for > 1 month (except for medications that will not affect the safety of the study and are not expected to affect any outcome of the study, in the judgment of the principal investigator)
* Live within a 60 minute drive-time radius of the central monitoring location
* Willing to remain within a 120 minute drive-time radius of the central monitoring location throughout the study
* Have someone over 18 years of age who lives with them, has access to where they sleep, is willing to be in the house when the subject is sleeping, and is willing to receive calls from the study staff and check the welfare of the study subject if telemetry shows a technical problem or severe biochemical hypoglycemia without subject response and the subject does not answer their telephone (up to two individuals can share this role, but they must be willing to carefully coordinate with each other and the subject so that one of them is clearly designated as having this responsibility at any given time)
* Willing to wear two infusion sets and one CGM sensor and change sets frequently (at least one new glucagon infusion set daily during bi-hormonal arms, and insulin infusion set every other day throughout the study)
* Have a mobile phone they are willing to keep with them and answer calls from study staff

Exclusion Criteria:

* Unable to provide informed consent (e.g. impaired cognition or judgment)
* Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory, unable to speak and read English)
* Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the subject
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception
* Need to go outside of the designated geographic boundaries during the study
* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days), use of marijuana within 1 month of enrollment, or other substance abuse (use within the last 6 months of controlled substances other than marijuana without a prescription)
* Unwilling or unable to refrain from drinking more than 2 drinks in an hour or more than 4 drinks in a day or use of marijuana during the trial
* Unwilling or unable or to avoid use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of beta blockers will be allowed as long as the dose is stable and the subject does not meet the criteria for hypoglycemia unawareness while taking that stable dose, but use of benzodiazepines or narcotics, even if by prescription, may be excluded according to the judgment of the principal investigator)
* History of liver disease that is expected to interfere with the anti-hypoglycemia action of glucagon (e.g. liver failure or cirrhosis). Other liver disease (i.e. active hepatitis, steatosis, active biliary disease, any tumor of the liver, hemochromatosis, glycogen storage disease) may exclude the subject if it causes significant compromise to liver function or may do so in an unpredictable fashion.
* Renal failure on dialysis
* Personal history of cystic fibrosis, pancreatitis, pancreatic tumor, or any other pancreatic disease besides type 1 diabetes
* Any known history of coronary artery disease including, but not limited to, history of myocardial infarction, stress test showing ischemia, history of angina, or history of intervention such as coronary artery bypass grafting, percutaneous coronary intervention, or enzymatic lysis of a presumed coronary occlusion)
* Abnormal EKG consistent with coronary artery disease or increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, prior myocardial infarction, proximal LAD critical stenosis (Wellen's sign), prolonged QT interval (> 440 ms). Non-specific ST segment and T wave changes are not grounds for exclusion in the absence of symptoms or history of heart disease. A reassuring evaluation by a cardiologist after an abnormal EKG finding may allow participation.
* Congestive heart failure (established history of CHF, lower extremity edema, paroxysmal nocturnal dyspnea, or orthopnea)
* History of TIA or stroke
* Seizure disorder, history of any non-hypoglycemic seizure within the last two years, or ongoing treatment with anticonvulsants
* History of hypoglycemic seizures (grand-mal) or coma in the last year
* History of pheochromocytoma: fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor:

oEpisodic or treatment refractory (requiring 4 or more medications to achieve normotension) hypertension oParoxysms of tachycardia, pallor, or headache oPersonal or family history of MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease

* History of adrenal disease or tumor
* Hypertension with systolic BP ≥160 mm Hg or diastolic BP ≥100 despite treatment
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
* Unable to completely avoid acetaminophen for duration of study
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study
* History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
* History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
* Type 1 diabetes subjects: Use of oral (e.g. thiazolidinediones, biguanides, sulfonylureas, glitinides, DPP-4 inhibitors, SGLT-2 inhibitors) anti-diabetic medications
* Type 2 diabetes subjects: Use of oral anti-diabetic medications other than metformin
* Lives in or frequents areas with poor Verizon wireless network coverage (which would prevent remote monitoring)
* Any factors that, in the opinion of the principal investigator would interfere with the safe completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Masscahusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.bionicpancreas.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 subjects were recruited and found eligible. Of the 27, only 24 subjects participated in the trial.
Pre-assignment Details: There were 24 subjects and a total of 9 study arms.The order of the arms was assigned in a psuedo random cross-over design. The 110 and 120 mg/dl arms were added later and were not included in the original randomization. 11 of the same subjects completed all 9 arms. Each arm had 20 subjects total, but these 20 were not the same cohort in each arm.
Groups:
- 110B, 110IO: Arms were completed in the following order: 110 mg/dl bihormonal bionic pancreas, 110 mg/dl insulin only bionic pancreas
- 110B, 110IO, 120IO: Arms were completed in the following order:
  110 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 120 mg/dl insulin only bionic pancreas
- 110IO, 110B, 120IO: Arms were completed in the following order: 110 mg/dl insulin only bionic pancreas, 110 mg/dl bihormonal bionic pancreas, 120 mg/dl insulin only bionic pancreas
- UC, 115B, 100B, 145IO, 130B, 130IO: Arms were completed in the following order: usual care, 115 mg/dl bihormonal bionic pancreas, 100 mg/dl bihormonal bionic pancreas, 145 mg/dl insulin only bionic pancreas, 130 mg/dl bihormonal bionic pancreas, 130 mg/dl insulin only bionic pancreas
- 145IO, 100B, 130B, 130IO, UC, 115: Arms were completed in the following order: 145 mg/dl insulin only bionic pancreas, 100 mg/dl bihormonal bionic pancreas, 130 mg/dl bihormonal bionic pancreas, 130 mg/dl insulin only bionic pancreas, usual care, 115 mg/dl bihormonal bionic pancreas
- UC, 115B, 145IO, 100B, 130IO, 130B: Arms were completed in the following order: usual care, 115 mg/dl bihormonal bionic pancreas, 145 mg/dl insulin only bionic pancreas, 100 mg/dl bihormonal bionic pancreas, 130 mg/dl insulin only bionic pancreas, 130 mg/dl bihormonal bionic pancreas
- 130B, 130IO, 115B, UC, 100B, 145IO, 120IO: Arms were completed in the following order: 130 mg/dl bihormonal bionic pancreas, 130 mg/dl insulin only bionic pancreas, 115 mg/dl bihormonal bionic pancreas, usual care, 100 mg/dl bihormonal bionic pancreas, 145 mg/dl insulin only bionic pancreas, 120 mg/dl insulin only bionic pancreas
- 145IO, 100B, UC, 115B, 130IO, 130B, 110B, 110IO: Arms were completed in the following order: 145 mg/dl insulin only bionic pancreas, 100 mg/dl bihormonal bionic pancreas, usual care, 115 mg/dl bihormonal bionic pancreas, 130 mg/dl insulin only bionic pancreas, 130 mg/dl bihormonal bionic pancreas, 110 mg/dl bihormonal bionic pancreas, 110 mg/dl insulin only bionic pancreas
- UC, 115B, 100B, 145IO, 130IO, 130B, 110IO, 110B: Arms were completed int he following order: usual care, 115 mg/dl bihormonal bionic pancreas, 100 mg/dl bihormonal bionic pancreas, 145 mg/dl insulin only bionic pancreas, 130 mg/dl insulin only bionic pancreas, 130 mg/dl bihormonal bionic pancreas, 110 mg/dl insulin only bionic pancreas, 110 mg/dl bihormonal bionic pancreas
- 130IO, 130B, UC, 145IO, 115B, 100B, 110B, 110IO: Arms were completed in the following order: 130 mg/dl insulin only bionic pancreas, 130 mg/dl bihormonal bionic pancreas, usual care, 145 mg/dl insulin only bionic pancreas, 115 mg/dl bihormonal bionic pancreas, 100 mg/dl bihormonal bionic pancreas, 110 mg/dl bihormonal bionic pancreas, 110 mg/dl insulin only bionic pancreas
- 130B, 130IO, UC, 145IO, 115B, 100B, 110B, 110IO: Arms were completed in the following order: 130 mg/dl bihormonal bionic pancreas,130 mg/dl insulin only bionic pancreas, usual care, 145 mg/dl insulin only bionic pancreas, 115 mg/dl bihormonal bionic pancreas, 100 mg/dl bihormonal bionic pancreas, 110 mg/dl insulin only bionic pancreas, 110 mg/dl bihormonal bionic pancreas
- 100B, 145IO, UC, 115B, 130IO, 130B, 110IO, 110B: Arms were completed in the following order: 100 mg/dl bihormonal bionic pancreas, 145 mg/dl insulin only bionic pancreas, usual care, 115 mg/dl bihormonal bionic pancreas, 130 mg/dl insulin only bionic pancreas, 130 mg/dl bihormonal bionic pancreas, 110 mg/dl insulin only bionic pancreas, 110 mg/dl bihormonal bionic pancreas
- 130IO, 130B, 145IO, 100B, 115B, UC, 110B, 110IO, 120IO: Arms were completed in the following order:
  130 mg/dl insulin only bionic pancreas 130 mg/dl bihormonal bionic pancreas 145 mg/dl insulin only bionic pancreas 100 mg/dl bihormonal bionic pancreas 115 mg/dl bihormonal bionic pancreas Usual Care 110 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 120 mg/dl insulin only bionic pancreas
- 115B, UC, 130B, 130IO, 145IO, 100B, 110IO, 110B, 120IO: Arms were completed in the following order:
  115 mg/dl bihormonal bionic pancreas Usual Care 130 mg/dl bihormonal bionic pancreas 130 mg/dl insulin only bionic pancreas 145 mg/dl insulin only bionic pancreas 100 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 110 mg/dl bihormonal bionic pancreas 120 mg/dl insulin only bionic pancreas
- UC, 145IO, 130B, 130IO, 100B, 115B, 110IO, 110B, 120IO: Arms were completed in the following order:
  Usual Care 145 mg/dl insulin only bionic pancreas 130 mg/dl bihormonal bionic pancreas 130 mg/dl insulin only bionic pancreas 100 mg/dl bihormonal bionic pancreas 115 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 110 mg/dl bihormonal bionic pancreas 120 mg/dl insulin only bionic pancreas
- UC, 145IO, 130B, 130IO, 100B, 115B, 110B, 110IO, 120IO: Arms were completed in the following order:
  Usual Care 145 mg/dl insulin only bionic pancreas 130 mg/dl bihormonal bionic pancreas 130 mg/dl insulin only bionic pancreas 100 mg/dl bihormonal bionic pancreas 115 mg/dl bihormonal bionic pancreas 110 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 120 mg/dl insulin only bionic pancreas
- 145IO, 100B, UC, 115B, 130B, 130IO, 110IO, 110B, 120IO: Arms were completed in the following order:
  145 mg/dl insulin only bionic pancreas 100 mg/dl bihormonal bionic pancreas Usual Care 115 mg/dl bihormonal bionic pancreas 130 mg/dl bihormonal bionic pancreas 130 mg/dl insulin only bionic pancreas 110 mg/dl insulin only bionic pancreas 110 mg/dl bihormonal bionic pancreas 120 mg/dl insulin only bionic pancreas
- 115B, UC, 130B, 130IO, 145IO, 100B, 110B, 110IO, 120IO: Arms were completed in the following order:
  115 mg/dl bihormonal bionic pancreas Usual Care 130 mg/dl bihormonal bionic pancreas 130 mg/dl insulin only bionic pancreas 145 mg/dl insulin only bionic pancreas 100 mg/dl bihormonal bionic pancreas 110 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 120 mg/dl insulin only bionic pancreas
- 130IO, 130B, 145IO, 100B, 115B, UC, 110IO, 110B, 120IO: Arms were completed in the following order:
  130 mg/dl insulin only bionic pancreas 130 mg/dl bihormonal bionic pancreas 145 mg/dl insulin only bionic pancreas 100 mg/dl bihormonal bionic pancreas 115 mg/dl bihormonal bionic pancreas Usual Care 110 mg/dl insulin only bionic pancreas 110 mg/dl bihormonal bionic pancreas 120 mg/dl insulin only bionic pancreas
- 100B, 145IO, UC, 115B, 130IO, 130B, 110IO, 110B, 120IO: Arms were completed in the following order:
  100 mg/dl bihormonal bionic pancreas 145 mg/dl insulin only bionic pancreas Usual Care 115 mg/dl bihormonal bionic pancreas 130 mg/dl insulin only bionic pancreas 130 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 110 mg/dl bihormonal bionic pancreas 120 mg/dl insulin only bionic pancreas
- UC, 115B, 145IO, 100B, 130B, 130IO, 110B, 110IO, 120: Arms were completed in the following order:
  Usual Care 115 mg/dl bihormonal bionic pancreas 145 mg/dl insulin only bionic pancreas 100 mg/dl bihormonal bionic pancreas 130 mg/dl bihormonal bionic pancreas 130 mg/dl insulin only bionic pancreas 110 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 120 mg/dl insulin only bionic pancreas
- 145IO, 100B, 130B, 130IO, UC, 115B, 110IO, 110B, 120IO: Arms were completed in the following order:
  145 mg/dl insulin only bionic pancreas 100 mg/dl bihormonal bionic pancreas 130 mg/dl bihormonal bionic pancreas 130 mg/dl insulin only bionic pancreas Usual Care 115 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 110 mg/dl bihormonal bionic pancreas 120 mg/dl insulin only bionic pancreas
- 130IO, 130B, 115B, UC, 100B, 145IO, 110B, 110IO, 120IO: Arms were completed in the following order:
  130 mg/dl insulin only bionic pancreas 130 mg/dl bihormonal bionic pancreas 115 mg/dl bihormonal bionic pancreas Usual Care 100 mg/dl bihormonal bionic pancreas 145 mg/dl insulin only bionic pancreas 110 mg/dl bihormonal bionic pancreas 110 mg/dl insulin only bionic pancreas 120 mg/dl insulin only bionic pancreas
Period: Overall Study
Arm/Group | 110B, 110IO | 110B, 110IO, 120IO | 110IO, 110B, 120IO | UC, 115B, 100B, 145IO, 130B, 130IO | 145IO, 100B, 130B, 130IO, UC, 115 | UC, 115B, 145IO, 100B, 130IO, 130B | 130B, 130IO, 115B, UC, 100B, 145IO, 120IO | 145IO, 100B, UC, 115B, 130IO, 130B, 110B, 110IO | UC, 115B, 100B, 145IO, 130IO, 130B, 110IO, 110B | 130IO, 130B, UC, 145IO, 115B, 100B, 110B, 110IO | 130B, 130IO, UC, 145IO, 115B, 100B, 110B, 110IO | 100B, 145IO, UC, 115B, 130IO, 130B, 110IO, 110B | 130IO, 130B, 145IO, 100B, 115B, UC, 110B, 110IO, 120IO | 115B, UC, 130B, 130IO, 145IO, 100B, 110IO, 110B, 120IO | UC, 145IO, 130B, 130IO, 100B, 115B, 110IO, 110B, 120IO | UC, 145IO, 130B, 130IO, 100B, 115B, 110B, 110IO, 120IO | 145IO, 100B, UC, 115B, 130B, 130IO, 110IO, 110B, 120IO | 115B, UC, 130B, 130IO, 145IO, 100B, 110B, 110IO, 120IO | 130IO, 130B, 145IO, 100B, 115B, UC, 110IO, 110B, 120IO | 100B, 145IO, UC, 115B, 130IO, 130B, 110IO, 110B, 120IO | UC, 115B, 145IO, 100B, 130B, 130IO, 110B, 110IO, 120 | 145IO, 100B, 130B, 130IO, UC, 115B, 110IO, 110B, 120IO | 130IO, 130B, 115B, UC, 100B, 145IO, 110B, 110IO, 120IO
Started | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 27 subjects were recruited and found eligible but 3 subjects chose not to participate in the study after eligibility determination
Groups:
- All Enrolled Subjects: All subjects enrolled into the study
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Hemoglobin A1c [Mean (Standard Deviation); unit: percent] | 7.3 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Continuous Glucose Monitor (CGM) Glucose Values
Description: Glucose values were collected from the Dexcom G4 CGM device every 5 minutes and an average (calculated mean with associated standard deviation) CGM glucose level (mg/dl) was calculated from days 2 and 3 of the study arm.
Time Frame: Days 2 and 3
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Usual Care | 145 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Bihormonal | 115 mg/dl Set Point - Bihormonal | 100 mg/dl Set Point - Bihormonal | 110 mg/dl Set Point - Insulin Only | 110 mg/dl Set Point - Bihormonal | 120 mg/dl Set Point - Insulin Only
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 14
mg/dl | 158 (31) | 174 (23) | 161 (17) | 156 (12) | 146 (15) | 136 (14) | 153 (15) | 148 (17) | 156 (15)

2. Primary Outcome: Percentage of Time With CGM < 60 mg/dl
Description: For this calculation we analyzed data from every 5 minutes of CGM data for days 2 and 3 of each study arm. We looked specifically at the percentage time of those roughly 48 hours that had any glucose values less than 60 mg/dl. The final value presented is the percent of time per 2 days of the study arm spent in a specific hypoglycemia range of less than 60 mg/dl with an associated standard deviation.
Time Frame: Days 2 and 3
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | 145 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Bihormonal | 115 mg/dl Set Point - Bihormonal | 100 mg/dl Set Point - Bihormonal | 110 mg/dl Set Point - Insulin Only | 110 mg/dl Set Point - Bihormonal | 120 mg/dl Set Point - Insulin Only
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 14
percentage of time | 1.38 (2.6) | 0.96 (1.5) | 0.79 (1.4) | 0.55 (1.0) | 0.88 (1.2) | 0.76 (1.1) | 1.34 (1.3) | 0.4 (0.6) | 1.05 (1.7)

3. Primary Outcome: Number of Subjects Discordant for Reaching a BG < 60 mg/dl for > 2 Consecutive Plasma Glucose Measurements During Inpatient Exercise Visit
Description: During both 110 mg/dl and 130 mg/dl arms, subjects will report for a fasted in-clinic exercise visit, with plasma blood glucose measurements obtained at least every 10 minutes
Time Frame: Day 4 in-clinic Exercise Visit (110 and 130 mg/dl arms only)
Measure: Count of Participants; unit: Participants
Groups:
- 130 mg/dl Insulin Only Bionic Pancreas: Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 130 mg/dl and using only an insulin pump. This arm is double blinded; neither the subject nor the study team know if it is insulin only or bihormonal.
- 130 mg/dl Bihormonal Bionic Pancreas: Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 130 mg/dl using both an insulin and a glucagon pump. This arm is double blinded; neither the subject nor the study team know if it is insulin only or bihormonal.
- 110 mg/dl Insulin Only Bionic Pancreas: Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 110 mg/dl and using only an insulin pump. This arm is double blinded; neither the subject nor the study team know if it is insulin only or bihormonal.
- 110 mg/dl Bihormonal Bionic Pancreas: Automated blood glucose control via a closed-loop bionic pancreas device targeting a blood glucose level of 110 mg/dl using both an insulin and a glucagon pump. This arm is double blinded; neither the subject nor the study team know if it is insulin only or bihormonal.
Arm/Group | 130 mg/dl Insulin Only Bionic Pancreas | 130 mg/dl Bihormonal Bionic Pancreas | 110 mg/dl Insulin Only Bionic Pancreas | 110 mg/dl Bihormonal Bionic Pancreas
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants | 0 | 0 | 3 | 1

4. Secondary Outcome: Mean CGM Glucose
Description: Average glucose according to continuous glucose monitor readings including the 1 day washout
Time Frame: Days 1 through 3
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Usual Care | 145 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Bihormonal | 115 mg/dl Set Point - Bihormonal | 100 mg/dl Set Point - Bihormonal | 110 mg/dl Set Point - Insulin Only | 110 mg/dl Set Point - Bihormonal | 120 mg/dl Set Point - Insulin Only
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 14
mg/dl | 160.8 (30.4) | 177.8 (19.5) | 164.1 (15.3) | 159.4 (13.4) | 151.6 (16.1) | 140.7 (15.4) | 158.8 (18.4) | 155.0 (19.4) | 160.2 (18.9)

5. Secondary Outcome: Nausea Severity
Description: The average severity of nausea, as recorded on a 10 centimeter visual analog scale by the daily e-mail survey they receive. Scores were determined by how many centimeters the subject marked as a surrogate for their nausea level on a daily basis. Any value more than 0 cm indicates some degree of nausea with a score of 10 cm being the worst nausea imaginable. A score less than 3 cm indicates a mild level of nausea.
Time Frame: Days 1-3
Measure: Mean (Standard Deviation); unit: scores on a scale 0-10 cm
Arm/Group | Usual Care | 145 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Bihormonal | 115 mg/dl Set Point - Bihormonal | 100 mg/dl Set Point - Bihormonal | 110 mg/dl Set Point - Insulin Only | 110 mg/dl Set Point - Bihormonal | 120 mg/dl Set Point - Insulin Only
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
scores on a scale 0-10 cm | 0.3 (0.5) | 0.5 (1.6) | 0.4 (0.6) | 0.4 (0.6) | 0.8 (1.6) | 1.2 (1.8) | 0.64 (1.25) | 0.80 (1.38) | 0.26 (0.26)

6. Secondary Outcome: Percentage of Time Spent in: < 50 mg/dl, < 70 mg/dl, 70-120 mg/dl, 70-180 mg/dl, > 180 mg/dl, >250 mg/dl
Description: The fraction of time spent in each of these ranges according to continuous glucose monitor readings
Time Frame: Days 2-3
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | 145 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Bihormonal | 115 mg/dl Set Point - Bihormonal | 100 mg/dl Set Point - Bihormonal | 110 mg/dl Set Point - Insulin Only | 110 mg/dl Set Point - Bihormonal | 120 mg/dl Set Point - Insulin Only
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 14
percentage of time
  < 50 mg/dl | 0.3 (0.6) | 0.5 (1.0) | 0.2 (0.8) | 0.1 (0.3) | 0.2 (0.4) | 0.2 (0.7) | 0.5 (0.7) | 0.1 (0.2) | 0.3 (0.6)
  < 70 mg/dl | 3.8 (6.2) | 2.4 (2.2) | 2.3 (2.1) | 1.3 (2.0) | 2.3 (2.3) | 2.4 (2.0) | 3.6 (2.2) | 1.2 (1.3) | 2.4 (3.3)
  70-120 mg/dl | 29.3 (18.8) | 16.9 (5.8) | 21.3 (7.4) | 25.9 (10.2) | 34.3 (8.2) | 45.3 (11.1) | 30.2 (7.1) | 37.5 (10.5) | 25.1 (7.6)
  70-180 mg/dl | 62.5 (19.0) | 57.0 (11.2) | 67.2 (13.6) | 70.8 (10.2) | 76.1 (11.0) | 80.7 (8.2) | 70.4 (10.3) | 76.5 (11.2) | 69.5 (14.0)
  > 180 mg/dl | 33.7 (21.5) | 40.6 (40.9) | 30.5 (13.1) | 27.9 (9.8) | 21.6 (10.3) | 16.9 (8.5) | 26.0 (10.2) | 22.2 (11.6) | 28.2 (12.9)
  > 250 mg/dl | 8.2 (8.4) | 11.3 (12.0) | 6.6 (7.3) | 5.1 (3.8) | 5.7 (6.7) | 3.4 (4.5) | 7.7 (6.2) | 6.5 (7.0) | 5.6 (6.0)

7. Secondary Outcome: Percentage of Subjects With Mean CGM < 154 mg/dl
Description: The percentage of subjects who's mean CGM glucose level is < 154 mg/dl, which is an estimated hemoglobin a1c < 7%, which is the ADA goal for therapy
Time Frame: Days 2-3
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | 145 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Insulin Only | 130 mg/dl Set Point - Bihormonal | 115 mg/dl Set Point - Bihormonal | 100 mg/dl Set Point - Bihormonal | 110 mg/dl Set Point - Insulin Only | 110 mg/dl Set Point - Bihormonal | 120 mg/dl Set Point - Insulin Only
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 14
Participants | 7 | 1 | 7 | 6 | 16 | 18 | 12 | 13 | 5

8. Secondary Outcome: Area Between the Glucose Curve and 60 mg/dl Calculated From BG Measurements
Description: Plasma glucose values to create this curve included time points from time 0 to a maximum of 360 minutes, with a sampling frequency of at least every 10 minutes throughout.
Time Frame: Day 4 in-clinic Exercise Visit (110 and 130 mg/dl arms only)
Measure: Mean (Standard Deviation); unit: min*mg/dl
Arm/Group | 130 mg/dl Insulin Only Bionic Pancreas | 130 mg/dl Bihormonal Bionic Pancreas | 110 mg/dl Insulin Only Bionic Pancreas | 110 mg/dl Bihormonal Bionic Pancreas
Number analyzed (Participants) | 20 | 20 | 20 | 20
min*mg/dl | 0 (0) | 0 (0) | 26.3 (78.5) | 5.15 (23.03)

9. Secondary Outcome: Area Between the Glucose Curve and 60 mg/dl Calculated From CGM Measurements
Description: CGM glucose values to create this curve included time points from time 0 to a maximum of 360 minutes, with a sampling frequency of every 5 minutes
Time Frame: Day 4 in-clinic Exercise Visit (type 1 diabetes only, 110 and 130 mg/dl arms only)
Measure: Mean (Standard Deviation); unit: min*mg/dl
Arm/Group | 130 mg/dl Insulin Only Bionic Pancreas | 130 mg/dl Bihormonal Bionic Pancreas | 110 mg/dl Insulin Only Bionic Pancreas | 110 mg/dl Bihormonal Bionic Pancreas
Number analyzed (Participants) | 20 | 20 | 20 | 20
min*mg/dl | 14.8 (66.2) | 0 (0) | 29.6 (91.5) | 0 (0)

10. Secondary Outcome: Time From Start of Exercise to First BG Measurement < 60 mg/dl
Description: as for outcome 3
Time Frame: Day 4 in-clinic Exercise Visit (type 1 diabetes only, 110 and 130 mg/dl arms only)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 130 mg/dl Insulin Only Bionic Pancreas | 130 mg/dl Bihormonal Bionic Pancreas | 110 mg/dl Insulin Only Bionic Pancreas | 110 mg/dl Bihormonal Bionic Pancreas
Number analyzed (Participants) | 20 | 20 | 20 | 20
minutes | NA (NA) — No BG values < 60 were reached during 130 arms | NA (NA) — No BG values < 60 were reached during 130 arms | 46.7 (59.2) | 30 (0)

11. Secondary Outcome: Time From Start of Exercise to First CGM Measurement < 60 mg/dl
Description: as for outcome 3
Time Frame: Day 4 in-clinic Exercise Visit (110 and 130 mg/dl arms only)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 130 mg/dl Insulin Only Bionic Pancreas | 130 mg/dl Bihormonal Bionic Pancreas | 110 mg/dl Insulin Only Bionic Pancreas | 110 mg/dl Bihormonal Bionic Pancreas
Number analyzed (Participants) | 20 | 20 | 20 | 20
minutes | 25.0 (0) | NA (NA) — There were no CGM values < 60 mg/dl in this arm | 53.3 (31.7) | NA (NA) — There were no CGM values < 60 mg/dl in this arm

12. Secondary Outcome: Grams of Carbohydrates Given to the Subject to Treat Hypoglycemia
Description: as for outcome 3
Time Frame: Day 4 in-clinic Exercise Visit (110 and 130 mg/dl arms only)
Measure: Mean (Standard Deviation); unit: grams of carbohydrates
Arm/Group | 130 mg/dl Insulin Only Bionic Pancreas | 130 mg/dl Bihormonal Bionic Pancreas | 110 mg/dl Insulin Only Bionic Pancreas | 110 mg/dl Bihormonal Bionic Pancreas
Number analyzed (Participants) | 20 | 20 | 20 | 20
grams of carbohydrates | 0 (0) | 0 (0) | 1.77 (5.51) | 0.86 (3.83)

13. Secondary Outcome: Total Glucagon Dosing by the Bihormonal Bionic Pancreas From the Start of Exercise Until the End of the Visit
Description: as for outcome 3
Time Frame: Day 4 in-clinic Exercise Visit (110 and 130 mg/dl arms only)
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | 130 mg/dl Insulin Only Bionic Pancreas | 130 mg/dl Bihormonal Bionic Pancreas | 110 mg/dl Insulin Only Bionic Pancreas | 110 mg/dl Bihormonal Bionic Pancreas
Number analyzed (Participants) | 20 | 20 | 20 | 20
mcg/kg | 0.0 (0.0) | 1.36 (1.06) | 0.0 (0.0) | 0.70 (0.53)

ADVERSE EVENTS:
Time Frame: Days 1-3 of each study arm
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT02509065/Prot_SAP_000.pdf